CLINICAL TRIAL: NCT06251583
Title: Prevention of Incisional Hernia With Mesh-suture (Duramesh Suture) at Umbilical Trocar Site in Patients Who Undergo Laparoscopic Surgical Approach
Brief Title: Prevention of Incisional Hernia With Mesh-suture at Umbilical Trocar Site.
Acronym: INDURATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Miguel A ngel Garci-a Urena (Other)
Collaborators: Ana Sánchez Gollarte (Unknown); Álvaro Robin Valle de Lersundi (Unknown); Arturo Cruz Cidoncha (Unknown); Almudena Moreno Elola-Olaso (Unknown); Armando Galván Pérez (Unknown); Ana María Minaya Bravo (Unknown); Enrique González González (Unknown); Carlos Guijarro Moreno (Unknown); Asunción Aguilera Velardo (Unknown); Patricia López Quindos (Unknown); Clara María Martínez Moreno (Unknown); Marina Pérez-Flecha González (Unknown); Victor Vaello Jodra (Unknown)
Responsible Party: Sponsor-Investigator, Miguel A ngel Garci-a Urena, Professor Miguel Ángel García Ureña, Henares University Hospital
Organization: Henares University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: INDURATE
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Incisional Hernia of Anterior Abdominal Wall; Dehiscence Wound; Wound Infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental group or Duramesh group (Experimental): Umbilical trocar closure using Suture-mesh (Duramesh suture).
  Interventions: Device: duramesh suture
- Control group or poli(4)hidroxibutirate group (Active Comparator): Umbilical trocar closure using conventional monofilament suture.
  Interventions: Device: duramesh suture

INTERVENTIONS:
Device: duramesh suture — Duramesh-suture will be used for trocar closure in the experimental group

SUMMARY:
Incisional hernia related to the umbilical trocar site is probably the most frequent complication after laparoscopic surgical procedures. However, this is an underestimated sequelae of laparoscopic surgery which may involve an important morbidity and an increase in healthcare costs.

The incidence of incisional trocar site hernia ranges from 20 to 35% of patients after laparoscopic surgery depending on the different investigations. Prophylactic meshes have been tried in an attempt to reduce the incidence of this complication in obese patients. In that sense, suture-meshes can be an alternative to conventional meshes to improve the incidence of incisional hernias.

INDURATE TRIAL aims to test if suture-mesh is capable of reducing the incidence of incisional hernia in patients with risk factors for the development of this frequent complication when compared with conventional monofilament sutures.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 year-old patients)
* Umbilical trocar incision > 10 mm
* Any of the following risk factors: BMI > 27, Absence of primary umbilical hernia or smaller than 1 cm, active smoking, malnutrition, anemia, oncological surgery, diabetes, heart failure, chronic kidney disease, chronic liver disease, collagen disease, chronic pulmonary disease.

Exclusion Criteria:

* Umbilical trocar incision < 10 mm
* Umbilical hernia > 10 mm
* Hernia surgery or incisional hernia at the trocar site
* Conversion to laparotomy
* Pregnancy
* Ascites or cirrhosis
* Clasification of the American Anestesiology Classification IV o V.
* Inadequate follow-up
* Patients included in any other trial
* Patients with life expectancy < 12 months
* Patients with any kind of sensibility to Duramesh

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-03-22 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of the umbilical trocar site hernia in each group | 12 monts
  Evaluation of the incidence of umbilical trocar site hernia in duramesh group compared with the control group

SECONDARY OUTCOMES:
Infectious complications of the wound | 12 months
  Evaluation of the infectious complications related to umbilical wound after laparoscopic surgery. Compare the incidence of these complications in each group
Seroma and hematoma | 12 months
  Evaluation of the seroma and hematoma related to umbilical wound after laparoscopic surgery. Compare the incidence of these complications in each group
Intraabdominal events | 12 months
  Evaluation of intraabdominal events (fluid collections, bleeding, peritonitis...) and compare the incidence in each group.
Skin dehiscence and/or necrosis | 12 months
  Evaluate the incidence of skin complications in each group.
Early aponeurotic failure (evisceration) | 12 months
  Evaluation of early aponeurotic failure after laparoscopic procuderes and compare the incidence between the two different groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Ángel García Ureña, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided